CLINICAL TRIAL: NCT01100008
Title: Cardiac Magnetic Resonance Imaging and Pulmonary Perfusion: Its Role in the Diagnosis of the Severity of Pulmonary Hypertension in Adults and in the Follow-up. Preliminary Study.
Brief Title: Cardiac Magnetic Resonance Imaging and Pulmonary Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06 042 02
Record Dates: First submitted 2010-03-01; First posted 2010-04-08 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary arterial hypertension; cardiac MRI (magnetic resonance imaging); severity; prognosis
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic resonance imaging (Experimental)
  Interventions: Procedure: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Procedure: Magnetic resonance imaging (MRI) — MRI cardiac and pulmonary with gadolinium

SUMMARY:
Pulmonary hypertension is a rare severe disease leading to cardiac insufficiency. Treatment depends on the severity of the disease.

This study evaluates cardiac MRI for the assessment of pulmonary hypertension severity and identification of parameters useful for the follow-up in order to adapt the medical treatment to status of the patient.

Evaluate if cardiac MRI can obviate right cardiac catheterization in the follow-up.

DETAILED DESCRIPTION:
Thirty patients will be enrolled and followed for 1 year after their inclusion.

Cardiac MRI will be performed at inclusion and at 3 months and 12 months. At the same periods, echocardiography and right heart catheterization will be performed too.

Morphological and functional parameters will be studied with MRI and correlated to invasive parameters and echocardiography too.

Morphological parameters are: volumes, cardiac cavities areas and ratios and position of the interventricular septum. Functional parameters are: ejection fractions of right and left cavities, flow in pulmonary artery, across mitral and tricuspid valves, temporal measurements in the pulmonary artery and auriculoventricular valves.

The invasive measurements are considered as the gold standard for this study. The classification of the severity is defined according to the parameters from right cardiac catheterization (4 grades with severity increasing between 1 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with pulmonary hypertension without specific treatment at inclusion
* Etiologies include chronic embolic disease, systemic fibrosis, Gougerot Sjogren, drug induced hypertension, primary hypertension.
* informed consent
* affiliated to medical insurance.

Exclusion Criteria:

* Left cardiac disease responsible for pulmonary hypertension, congenital cardiopathies
* Pulmonary functional tests with important impairment (decrease in TPCmore than 30%, decrease In VEMS more than 30%
* Child
* pregnancy
* contraindications to MRI
* without informed consent
* without insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-09; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Nuclear magnetic resonance imaging | Inclusion ; 3rd month ; 12th month
  Correlation of cardiac results from the first MRI (Magnetic Resonance Imaging) to invasive measurements from the first or initial right heart catheterization and to echocardiography to know if cardiac MRI is able to predict severity of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Chabbert, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Service de radiologie - Hôpital Rangueil, Toulouse, Midi-Pyrénées, France

IPD SHARING:
Plan to Share IPD: No